CLINICAL TRIAL: NCT07390032
Title: The Efficacy and Safety of Endovascular Treatment for Acute Mild Basilar Artery Occlusion: A Multicenter, Prospective, Open-Label, Endpoint-Blinded, Randomized Controlled Clinical Trial
Brief Title: The Efficacy and Safety of Endovascular Treatment for Acute Mild Basilar Artery Occlusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Feng Gao (Other)
Responsible Party: Sponsor-Investigator, Feng Gao, Vice-Director of Interventional Neuroradiology, Department of Neurology, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-A-2025111
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Acute Mild Basilar Artery Occlusion; Basilar Artery Occlusion; Endovascular Treatment
Keywords: Acute Ischemic Stroke; Acute Mild Basilar Artery Occlusion; Basilar Artery Occlusion; Endovascular Treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular Treatment Group (Experimental): Participants randomized to the endovascular recanalization arm will receive endovascular treatment in addition to best medical management. The procedure aims to achieve recanalization of the occluded basilar artery using mechanical thrombectomy techniques, including stent retriever and/or aspiration-based approaches. When necessary, adjunctive endovascular measures may be performed as rescue therapy at the discretion of the treating neurointerventionalist.
  Interventions: Procedure: Endovascular Recanalization Strategy
- Best Medical Management Group (Experimental): Participants randomized to this arm will receive best medical management alone, consistent with current guideline recommendations for the acute and secondary prevention phases of ischemic stroke. No endovascular recanalization procedures are permitted after randomization.
  Interventions: Drug: Best Medical Management

INTERVENTIONS:
Procedure: Endovascular Recanalization Strategy — The endovascular approach is selected by the treating neurointerventionalist based on angiographic findings, occlusion characteristics, and procedural feasibility. Permitted techniques include mechanical thrombectomy using stent retriever and/or aspiration-based methods. Adjunctive endovascular procedures, such as balloon angioplasty, stent placement, or intra-arterial thrombolysis, may be used when deemed necessary to achieve or maintain vessel patency. Angiographic reperfusion is assessed during the procedure, and treatment is terminated once adequate revascularization is obtained. Subsequent medical management is individualized according to stroke mechanism, procedural findings, and post-treatment imaging.
  Arms: Endovascular Treatment Group
Drug: Best Medical Management — Best medical management consists of comprehensive evidence-based medical therapy for acute ischemic stroke, encompassing acute supportive care, neurological and physiological monitoring, etiological evaluation, and secondary prevention strategies. Standard pharmacological treatments are administered as appropriate, together with risk factor modification and supportive care measures, in accordance with current guideline recommendations. Endovascular recanalization procedures are not included in this treatment strategy.
  Arms: Best Medical Management Group

SUMMARY:
This study assesses the efficacy and safety of endovascular treatment for acute mild basilar artery occlusion within a multicenter, prospective, open-label, endpoint-blinded, randomized controlled clinical trial.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, open-label, controlled trial with blinded outcome assessment (PROBE design) evaluating endovascular therapy (EVT) for patients with acute mild basilar artery occlusion (MBAO). Acute MBAO is defined as basilar artery occlusion confirmed by CTA/MRA/DSA, with mild neurological deficits (baseline NIHSS ≥2 and <10). Participants will be randomized in a 1:1 ratio to receive either EVT plus best medical therapy or best medical therapy alone. The primary outcome is the rate of good functional status at 90 days after randomization was defined as the modified Rankin Scale (mRS) score of 0-2 at 90 days. Secondary outcomes include the distribution of mRS scores at 90 days, 90-day all-cause mortality, and the incidence of symptomatic intracranial hemorrhage (sICH).

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18
2. Acute ischemic stroke in posterior circulation, the time from stroke onset (or finally found normal) to randomization was within 24 hours
3. Acute basilar artery occlusion confirmed by CTA,MRA,or DSA
4. NIHSS score≥2 points and<10 points from the onset of the disease to before randomization
5. Posterior circulation large core infarction:NCCT or DWI showed pc-ASPECTS≥6, or Pons-Midbrain Index (PMI)<3
6. No significant functional disability before stroke (mRS≤2 points)
7. Each patient or their legal representative must provide written informed consent before enrolment

Exclusion Criteria:

1. Any sign of intracranial hemorrhage (except microbleeds) on brain imaging prior to randomization
2. Complete cerebellar infarct with significant mass effect, or bilateral thalamic infarction as evidenced by baseline neuroimaging
3. Known or highly suspected chronic occlusion of basilar artery
4. History of contraindication for contrast medium (except mild rash)
5. CTA/MRA/DSA confirmed occlusion of anterior and posterior circulation
6. Severe stenosis, arterial dissection, or excessive tortuosity of the extracranial or intracranial segments of the vertebral artery may result in the inability of interventional instruments to be successfully delivered or positioned
7. Current pregnant or breast-feeding
8. Refractory hypertension (defined as systolic blood pressure>185 mmHg or diastolic blood pressure>110 mmHg) that cannot be controlled by drug treatment
9. Known hereditary or acquired bleeding tendency, lack of coagulation factors, or oral anticoagulants with INR>1.5
10. Blood glucose<2.8 or>22.2 mmol/L; Platelet count<100*109/L, serum creatinine>2.0 g/L (177 μ mol/L), or glomerular filtration rate<30 ml/(min*1.73 m2)
11. Enrolled in another drug or device trial or expected to participate in another drug or device treatment trial within the following 3 months
12. Acute cerebral infarction occurred within 48 hours after cardio cerebral vascular intervention or major surgery (patients over 48 hours can be included in the group)
13. Patients whose life expectancy is less than 1 year (such as patients with malignant tumor, advanced cardiopulmonary disease, etc.)
14. Central nervous system vasculitis has been diagnosed or clinically suspected
15. Known to have dementia or psychiatric disease unable to complete neurological assessment and follow-up
16. It is known that patients with dementia or mental illness cannot complete neurological function assessment and follow-up
17. Any other condition (in the opinion of the site investigator) that inappropriate to participate this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate modified Rankin Scale (mRS) score 0-2 at 90 days | 90±14 days after randomization
  The modified Rankin scale (mRS) ranged from 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability,5 severe disability, and 6 death.

SECONDARY OUTCOMES:
mRS score as an ordinal scale at 90 days after randomization | 90±14 days after randomization
  The modified Rankin scale (mRS) ranged from 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death.
The rate of 0-1 and 0-3 mRS scores after randomization for 90 days | 90±14 days after randomization
  The modified Rankin scale (mRS) ranged from 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death.
National Institutes of Health Stroke Scale (NIHSS) score at 24 hours after randomization | 24 (-6/+12) hours after randomization
  National Institutes of Health Stroke Scale (NIHSS) score at 24 hours after randomization The National Institute of Health Stroke Scale (NIHSS) ranged from 0 to 42, with higher scores indicating greater neurologic deficits.
NIHSS score at 7 days after randomization or discharge (whichever occurs first), as well as changes from baseline | 7 days after randomization or at discharge
  NIHSS score at 7 days after randomization or discharge (whichever came first) The National Institute of Health Stroke Scale (NIHSS) ranged from 0 to 42, with higher scores indicating greater neurologic deficits.
European Five Dimensional Health Scale Level 5 (EQ-5D-5L) score 90 days after randomization | 90±14 days after randomization
  EuroQol Five Dimensions (EQ-5D-5L) is a standardized instrument for measuring the general health status. Rated level can be coded as a number 1, 2, 3, 4 or 5, which indicates having no problems for 1, having some problems for 2, having moderate problems for 3, having serious problems for 4 and having extreme problems for 5.
Barthel index 95-100 points 90 days after randomization | 90±14 days after randomization
  The proportion of Barthel Index 95-100 at 90 days after randomization.
The recanalization of the basilar artery 24 hours after randomization (confirmed by CTA, MRA, DSA, or TCD) | 24 (-6/+12) hours after randomization
  Basilar artery recanalization at 24 hours after randomization (confirmed by CTA, MRA, DSA or TCD).
The technical success rate is defined as the successful recanalization of the target vessel at the end of the surgery (Extended Thrombolysis Classification for Cerebral Infarction [eTICI] 2b-3) | At the end of the operation
  Technical success rate, defined as successful recanalization of target vessels at the end of surgery (The expanded Thrombolysis in Cerebral Infarction (eTICI) scale eTICI 2b-3).

OTHER OUTCOMES:
Mortality rate within 90 days after randomization | 90±14 days after randomization
  All cause of mortality within 90 days after randomization.
Rate of any Symptomatic intracranial hemorrhage (sICH) defined as the Heidelberg classification within 24 hours of randomization | 24 (-6/+12) hours after randomization
  Heidelberg standard was defined as new intracranial hemorrhage detected by brain imaging associated with any of the item below: 4 points total NIHSS at the time of diagnosis compared to immediately before worsening. 2 point in one NIHSS category. Leading to intubation/hemicraniectomy/ventricular drainage placement or other major medical/surgical intervention. Absence of alternative explanation for deterioration.
Rate of any intracranial hemorrhage identified by CT or MRI imaging within 24 hours after randomization | 24 hours after randomization
  Any intracranial hemorrhage identified by CT or MRI imaging within 24 hours.
All cause of mortality within 7 days after randomization | 7 days after randomization or at discharge
  All cause of mortality within 7 days after randomization.
Surgical related complications: arterial perforation, arterial dissection, and embolism in newly developed vascular areas | At the end of the operation or intraoperative
  Surgical related complications: arterial perforation, arterial dissection, and embolism in newly developed vascular areas.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Gao, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No